CLINICAL TRIAL: NCT04599166
Title: Choosing an Effective Healthcare Spokesperson: An Interactive Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Benjamin H. Levi, Co-Principal Investigator, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IR-16274; R21NR019363 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Surrogate Decision-making; Healthcare Spokesperson; Advance Care Planning
Keywords: Surrogate decision-making; Healthcare spokesperson; Advance care planning; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant arm (Experimental): Participants will be recruited to complete the WWYC intervention.
  Interventions: Behavioral: Who Would You Choose: Serious Fun

INTERVENTIONS:
Behavioral: Who Would You Choose: Serious Fun — "Who Would You Choose: Serious Fun" is a conversation activity that prompts players (using scenarios and metaphors) to choose a spokesperson whose qualities are best suited to the role. At the end of the activity, players identify a real-life spokesperson based on the qualities considered during gameplay.

SUMMARY:
The investigators developed a "serious game" intervention called "Who Would You Choose: Serious Fun" (WWYC) to help people consider the key qualities healthcare spokespersons should have. The intervention uses a spinner, cards, and dice, along with a smart-phone App to prompt players (using scenarios and metaphors) to choose a spokesperson whose qualities are best suited to the role. Friendly competition is encouraged by having players receive points for correct answers, and additional points for good explanations of their choices. At the end of the game, players identify a real-life spokesperson based on the qualities considered during game-play. Then, using an associated smart-phone App, the intervention will help spark communication between the player and their chosen spokesperson.

DETAILED DESCRIPTION:
Advance care planning (ACP) is the process of thinking through and articulating in advance one's preferences for future medical care. It has long been promoted as a way for people to receive medical treatment consistent with their values, goals, and preferences. While ACP typically involves decision-making about specific life-sustaining treatments, choosing who will make medical decisions when the patient cannot is considered by many to be the single most important ACP action a person can take. When patients fail to designate a healthcare spokesperson (henceforth spokesperson), it leads to uncertainty about who will make medical decisions, what treatments are to be accepted or declined, and on what basis-which can lead to familial conflict, unwanted and costly medical care, and avoidable patient suffering. So, too, when patients choose the "wrong" person to represent them, the patient's wishes are less likely to be known or respected. The investigation team's own research suggests that when patients prefer fewer aggressive medical treatments, there is significantly lower concordance between spokespersons' decisions and patients' wishes.

Patients, families, and ACP experts have identified several qualities as being especially important for spokespersons to have. Ideally, spokespersons should know the patient's values, be available when needed, be trustworthy and caring, have good judgment, and be able to stand up under pressure. That said, many individuals (and state laws) assign spokespersons on the basis of relationship (spouse, parent, etc.) rather than personal qualities. Surprisingly, no interventions (to the team's knowledge) are explicitly designed to help people consider the actual qualities of the person chosen as spokesperson, much less engage this individual to confirm that this person can fully represent the patient's wishes should the need arise.

To address these gaps, the investigative team has developed a novel intervention that includes a "serious game" to help people consider the qualities desired in a spokesperson, then engage the person they choose for this role. Combining a serious topic with an enjoyable activity ("gamification") has been effective at changing health-related behaviors in multiple settings with the target population ("sandwich generation" and older adults). The game element of the intervention, "Who Would You Choose: Serious Fun" (WWYC), prompts players (using scenarios and metaphors) to choose a spokesperson whose qualities are best suited to the role. At the end of the game, players identify a real-life spokesperson based on the qualities considered during gameplay. Then, using an online interface, WWYC will spark communication between the player and their chosen spokesperson.

The long-term goal of this project is to help people make more thoughtful and informed choices when selecting a spokesperson, and to help these spokespersons be better prepared for the role of surrogate decision-maker. The current mixed methods study proposed here is designed to learn whether and how WWYC helps individuals select an appropriate spokesperson for healthcare decisions, as assessed via three specific aims:

Aim 1. To explore how playing the novel game Who Would You Choose affects people's choice of a spokesperson. Using qualitative methods including focus groups and one-on-one interviews, the investigative team will explore how WWYC affects individual players' thought process for choosing a spokesperson, and whether the player's choice changes as a result of game-play.

Aim 2. To establish that WWYC is a feasible way to help individuals choose and engage a spokesperson. The investigative team will judge it feasible if: 1) 100 individuals are recruited to play the game; 2) >75% of game players report that playing the game is helpful for choosing a spokesperson; 3) >75% of game players endorse the game; 4) >75% of spokespersons engage with WWYC (using its online interface) following player request.

Aim 3. To integrate qualitative and quantitative data to explain how the experience of playing the game relates to their spokesperson's willingness to engage. The investigative team hypothesizes that a positive player experience with WWYC will be associated with successful engagement with their spokesperson.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English
* 18 years or older
* Have a working smart phone

Exclusion Criteria:

* NOT able to read and write in English
* Younger than 18 years old
* Does NOT have a working smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Levi, MD PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will present our findings at conferences and in peer-reviewed publications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At close of study in 2022.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Flier, emails, and public service announcements were used to recruit community members for participation in study game events. Respondents were contacted via email and phone. A total of 207 individuals expressed interest and showed up to game events. The period of study recruitment was from 7-1-2020 - 11-1-2022.
Pre-assignment Details: Not applicable as there was only one arm to the study, and no participants were excluded after enrollment.
Groups:
- Participant Arm: Participants were recruited to complete the WWYC intervention.
  Who Would You Choose: Serious Fun: "Who Would You Choose: Serious Fun" is a conversation activity that prompts players (using scenarios and metaphors) to choose a spokesperson whose qualities are best suited to the role. At the end of the activity, players identify a real-life spokesperson based on the qualities considered during gameplay.
Period: Overall Study
Arm/Group | Participant Arm
Started | 207
Completed | 127
Not Completed | 80
Not completed — Technological failure connecting to study app | 80

BASELINE CHARACTERISTICS:
Arm/Group | Participant Arm
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (17)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 64
  Female | 58
  Other | 2
  Prefer not to answer | 1
  Missing data | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 15
  Asian | 11
  American Indian or Alaskan Native | 1
  Middle Eastern or North African | 0
  Native Hawaiian or Pacific Islander | 0
  White | 91
  Other | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127
Marital status [Count of Participants; unit: Participants]
  Missing | 1
  Single | 69
  Married | 43
  Divorced | 5
  Widowed | 3
  Civil Union/Domestic Partnership | 5
  Prefer not to answer | 1
Highest Level of Education [Count of Participants; unit: Participants]
  High school graduate | 9
  Trade or professional degree | 4
  Some college | 21
  Associate's degree | 13
  Bachelor's degree | 44
  Master's degree | 32
  Doctoral degree | 4
Healthcare worker status [Count of Participants; unit: Participants]
  Work in healthcare field | 16
  Do not work in healthcare field | 111
Prior experience with surrogate decision-making [Count of Participants; unit: Participants]
  Has made surrogate decision for another | 23
  Has not made surrogate decision for another | 104
Importance of religion or spirituality [Count of Participants; unit: Participants]
  Not at all important | 25
  Not very important | 24
  Somewhat important | 35
  Very important | 26
  Extremely important | 17
Health status [Count of Participants; unit: Participants]
  Excellent | 15
  Very good | 61
  Good | 42
  Fair | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Changed Their Choice of Spokesperson
Description: This measure involved a verbal response (during a follow-up telephone interview) to the question as to whether they have changed their choice for who should be their healthcare spokesperson in the event that someone else needed to make medical decisions for them.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Participant Arm: This was a 1-armed study in which all participants were asked to identify a real-life spokesperson after completing the intervention.
Arm/Group | Participant Arm
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Participation Rate
Description: Participation rate was defined as the number of participants who completed the study. This number excludes the number of participants who were enrolled but could not complete the intervention due to problems with technology (n=80).
Time Frame: Aug 2021 - Dec 2022
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Arm
Number analyzed (Participants) | 127
Participants | 127

3. Secondary Outcome: Spokesperson Response (Percentage)
Description: Percentage of spokespersons who responded to participant request following intervention
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Arm
Number analyzed (Participants) | 127
Participants
  Spokespersons who responded to invitation | 40
  Spokespersons who did not respond to invitation | 87

4. Secondary Outcome: Endorsement of the WWYC Intervention
Description: >75% of WWYC participants endorse WWYC, as measured by the Net Promoter Score
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Arm
Number analyzed (Participants) | 127
Participants | 97

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Participant Arm
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

LIMITATIONS AND CAVEATS:
1. At several game events, we experienced technology failures when participants tried to connect to the intervention app. This resulted in several events being cancelled, with no data collection from them.
2. We were unable to retrieve audio-recordings for one-on-one telephone interviews from the digital recording device, and are unable to report those qualitative data. This is why we only had results from 8 participants for the primary outcome of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT04599166/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04599166/ICF_001.pdf